CLINICAL TRIAL: NCT04061629
Title: Minimal Occlusive Pressure With Cuffed ETTs: The Effect of 3 Different Sizes of cETT on Intracuff Pressure in Children
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Senthil G. Krishna, Clinical Associate Professor of Anesthesiology, Nationwide Children's Hospital
Other Study IDs: IRB17-00700
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Surgical Procedure, Unspecified

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group C: Size of the cuffed ETT based on the Cole formula = (Age/4) + 4.
  Interventions: Device: Cuffed ETT
- Group D: size of the cuffed ETT based on the Duracher formula = (Age/4) + 3 + 0.5 mm.
  Interventions: Device: Cuffed ETT
- Group K: size of the cuffed ETT based on the Khine formula = (Age/4) + 3.
  Interventions: Device: Cuffed ETT

INTERVENTIONS:
Device: Cuffed ETT — Cuffed endotracheal tube.

SUMMARY:
Based on standard and historical practice, the predictive size of the endotracheal tube (ETT) to be used in children has been based on various formulas. However, no study has clearly compared these formulas to determine the optimal size of cuffed ETTs. Furthermore, they were developed when using a polyvinylchloride cuff and not the thinner polyurethane cuff which is in common clinical use today. Hence, the purpose of this current study is to evaluate which of the currently available formulas most closely predicts the appropriate size of cuffed ETT to be used based not only on the fit within the trachea, but more importantly the intracuff pressure after the cuff is inflated to seal the airway.

ELIGIBILITY:
Inclusion Criteria:

* Children who are less than 8 years of age and are scheduled for surgical procedures requiring endotracheal intubation with a cuffed ETT.

Exclusion Criteria:

* Children with airway anomalies or other factors that may impact tracheal size will be excluded from the study.

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children requiring an endotracheal tube for surgery.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Number of participants that needed their ETT exchanged | Immediately following intubation
  Having to remove the original ETT and replacing it with a smaller or larger size due to excessive air leak or excessive pressure in the cuff.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States